CLINICAL TRIAL: NCT06014203
Title: Examination of Edema After Arthroscopic Shoulder Surgery
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: Iayas5
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Edema; Arthroscopy; Shoulder
Keywords: Edema; Shoulder arthroscopy
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing shoulder arthroscopy surgery: Patients who underwent arthroscopic shoulder surgery by a single surgeon at Gazi Hospital Department of Orthopedics and Traumatology (rotator cuff repair, slap, bankart repair)
  Interventions: Diagnostic Test: Edema measurement

INTERVENTIONS:
Diagnostic Test: Edema measurement — Subcutaneous fluid measurements will be made 3 times in total, before the surgery, immediately after the surgery and 24 hours after the surgery. Measurements will be made with the MoistureMeterD Compact local edema measuring device.
  Points to be measured:
  1. Midpoint of the upper trapezius muscle
  2. 5 cm distal to anterior acromion
  3. 5cm distal to lateral acromion
  4. 5cm distal to posterior acromion
  5. 3cm medial to the axilla
  6. Anterior cubital fossa
  7. Carpal tunnel

SUMMARY:
The investigators's aim is to examine trunk and upper extremity edema after arthroscopic rotator cuff repair and/or labrum repair surgeries. During surgery, the shoulder joint capsule is cut and the joint is entered arthroscopically. During this procedure, approximately 3-6 liters of saline fluid is injected into the joint, depending on the duration of the surgery. The given fluid accumulates out of the joint in relation to the duration of the surgery and the amount of fluid given. In this study, the investigators aim is to examine how much the extra-articular fluid collects under the skin of the upper extremity and trunk, and the change in the amount of fluid 24 hours after surgery. Examination of the amount of subcutaneous fluid may help to better understand the postoperative complications such as edema, carpal tunnel syndrome, compartment syndrome, myolysis, and dyspnea. How much edema the joint and surrounding structures are exposed to and its relationship with the duration of surgery can help to clinicians determine the safe discharge time.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic shoulder surgery planned
* 18-65 years old

Exclusion Criteria:

* Frozen/stiff shoulder
* Metabolic and endocrine diseases
* Dermatological pathologies
* Hyperlaxity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for arthroscopic shoulder surgery in Gazi University Hospital, Department of Orthopedics and Traumatology
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Edema | 3 months
  After the MoistureMeterD Compact local edema measuring device is placed perpendicular to the area to be measured, it will be held for 3 seconds and the percent moisture value will be recorded. 3 measurements will be made for each region. The average of the 3 measurements will be used in the statistical analysis.

SECONDARY OUTCOMES:
Surgery time | 3 months
  The duration of each operation will be recorded in minutes by the surgeon performing the operation.
Amount of the saline | 3 months
  The amount of saline fluid used in each operation will be recorded in liters by the surgeon performing the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Ayas IH, Akcan YO, Haspolat M, Tokgoz MA, Keser I, Kanatli U. Subcutaneous Pectoral Edema After Arthroscopic Labral Repair Despite Normal Irrigation Fluid Usage and Surgery Duration. Orthop Surg. 2025 Feb;17(2):624-630. doi: 10.1111/os.14324. Epub 2025 Jan 15. PMID 39814377